CLINICAL TRIAL: NCT06003478
Title: The Safety and Influencing Factors of Ultrasound-guided Percutaneous Intramyocardial Septal Radiofrequency Ablation (Liwen Procedure) in The Treatment of Hypertrophic Cardiomyopathy
Brief Title: The Safety and Influencing Factors of Liwen Procedure in The Treatment of Hypertrophic Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Liu Liwen, Director, Xijing Hospital
Other Study IDs: KY20232228-C-1
Record Dates: First submitted 2023-08-11; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
Keywords: Cardiomyopathy, hypertrophic; Hypotension; Postoperative Complication
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypotension; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertrophic Obstructive Cardiomyopathy Patients
  Interventions: Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy (Liwen Procedure)

INTERVENTIONS:
Procedure: Percutaneous Intramyocardial Septal Radiofrequency Ablation for hypertrophic obstructive cardiomyopathy (Liwen Procedure) — Under transthoracic echocardiography (TTE) guidance, the puncture site is positioned at the apex. A guiding line is applied along the septal long axis and the radiofrequency ablation electrode needle(17G, Cool-tip™ RF Ablation System and Switching Controller;Medtronic, Minneapolis, MN, USA) pierced towards the hypertrophic anterior interventricular septum (AIVS) 8-10 mm from the subaortic valve. Each ablation lasts for up to 12 min and the ablation power is gradually increased from 30-40W. Then, the ablation needle is withdrawn 10 mm to prepare for the next application. Overall, 3-4 applications are performed in each patient. The ablation creates an area of thermal coagulative myocardial necrosis that appears as a hyperechogenic reflection detected by TTE. If deemed necessary, we repeat the procedure at the posterior interventricular septum (PIVS).

SUMMARY:
Liwen procedure is generally safe and effective in treating hypertrophic cardiomyopathy, but a small proportion of patients have complications after the operation.

The goal of this observational study is to explore the incidence of postoperative complications of the Liwen procedure in hypertrophic cardiomyopathy patients underwent Liwen procedure in Xijing Hospital. The main question it aims to answer are:

* What is the incidence of complications in HCM patients underwent Liwen Procedure during postoperative hospitalization and a short-term follow-up period?
* What is the relevant factors of complications in HCM patients who underwent Liwen Procedure during postoperative hospitalization and short-term follow-up period? Can the complications of surgical patients during postoperative hospitalization be predicted? Participants have been evaluated using a variety of medical examinations before they underwent Liwen Procedure. Variants collected from medical examination and case history were used to analyze the association with each postoperative complication.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with symptoms that limit daily activities (New York Heart Association functional class >II, exercise-induced syncope) despite adequate medical treatment or when medical treatment is not tolerated
2. Subject with a peak LVOT gradient≥50 mm Hg
3. Subject volunteers for the Liwen procedure and received the procedure at the Hypertrophic Cardiomyopathy Center of Xijing Hospital.

Exclusion Criteria:

1. Subject with a peak instantaneous Doppler LVOT gradient of <50 mm Hg
2. Subject with an indication for septal reduction therapy and other lesions requiring surgical intervention (e.g., mitral valve repair/replacement and papillary muscle intervention)
3. Subject has end-stage heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with obstructive HCM and with drug-refractory symptoms underwent Liwen Procedure in Xijing Hospital from 2016 October to 2023 July.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Complications During Hospitalization | From date of procedure until the date of first documented occurrence of symptomatic hypotension, or date of dischargement from hospital, assessed up to 1 month.
  Complications including symptomatic postoperative hypotension observed during hospitalization after PIMSRA. The symptomatic postoperative hypotension is defined as systolic blood pressure lower than 90 mmHg documented by invasive or noninvasive blood pressure measurement accompanied by symptoms including dizziness, and cephalalgia, without regard to the duration of hypotension.

SECONDARY OUTCOMES:
Postoperative Complications During Follow-up Period | From date of dischargement until the date of first diagnosis of chronic hypotension or orthostatic hypotension, assessed up to 1 year.
  Complications including chronic hypotension or orthostatic hypotension observed during the follow-up period. Chronic hypotension is defined as mean systolic/diastolic blood pressure lower than 90/60 mmHg documented by ambulatory blood pressure monitoring of more than 23 hours. Orthostatic hypotension is defined as a frop of standing and mean sitting SBP ≥20 mm Hg or diastolic BP ≥10 mm Hg, with complaining of dizziness or fall.

CONTACTS AND LOCATIONS:
Locations (1):
- Ultrasound Medicine Department of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Shan B, Li J, Shi Z, Han C, Zhang J, Zhao J, Hu R, Liu L, Ta S. Predictive value of estimated plasma volume for postoperative hypotension in percutaneous intramyocardial septal radiofrequency ablation treating for hypertrophic obstructive cardiomyopathy. BMC Cardiovasc Disord. 2024 Mar 22;24(1):177. doi: 10.1186/s12872-024-03844-9. PMID 38519968